CLINICAL TRIAL: NCT03077022
Title: Effectiveness of Physical Therapy (PT) Alone vs PT Followed by Surgery to Alleviate the Symptoms of Femoroacetabular Impingement (FAI)
Brief Title: Femoroacetabular Impingement (FAI): The Effectiveness of Physical Therapy
Status: Withdrawn | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-0244
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Femoracetabular impingent (FAI): Subjects will be given a prescription for physical therapy specifically for Femoracetabular impingent (FAI). They will then be followed clinically per the investigator's normal routine and the gold standard.

SUMMARY:
The treatment of femoroacetabular impingement has evolved over the last several years. As the number of arthroscopic hip operations has risen over the last few years, so has the level controversy in regards to the appropriate initial management. There have been many recent advances in clinical diagnosis, advanced imaging techniques, improved indications for surgery and improved arthroscopic techniques which have led to improved clinical outcomes, but the effectiveness of physical therapy remains unknown.

DETAILED DESCRIPTION:
The treatment of femoroacetabular impingement has evolved over the last several years. As the number of arthroscopic hip operations has risen over the last few years, so has the level controversy in regards to the appropriate initial management. There have been many recent advances in clinical diagnosis, advanced imaging techniques, improved indications for surgery and improved arthroscopic techniques which have led to improved clinical outcomes, but the effectiveness of physical therapy remains unknown.

A paucity of evidence exists in regards to the non-operative treatment of FAI.

Several insurance companies are now requiring three to six months of physical therapy prior to approval for surgery. There is not a single study that has objectively evaluated the effectiveness of physical therapy in the avoidance of surgical intervention. The investigators plan to evaluate this using an electronic outcomes data collection system. The hypothesis is that the majority of patients will not see a significant enough improvement with physical therapy to avoid surgery, especially in a subset of patients such as those with sub spine impingement. The investigators plan to prospectively collect data for three years and monitor the outcome of each hip patient, especially those treated with physical therapy as an initial treatment and there potential avoidance of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. symptoms consistent with femoroacetabular impingement (FAI)
2. a physical exam consistent with FAI
3. radiographic measurements consistent with the diagnosis including an anterior pincer lesion and/or a alpha angle greater than 55 degrees

Exclusion Criteria:

1. subjects do not have FAI by physical exam and radiographic parameters
2. joint space <2mm
3. have had prior physical therapy for FAI
4. have had prior hip surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be included if they are 18-65 years old. Patients with hip pain are routinely seen in our clinic. Patients who meet the inclusion/exclusion criteria will be offered the opportunity to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in sub spine impingement associated with physical therapy | Baseline, 6 weeks, 12 weeks, 3 months, 6 months, 1 year, and 2 years.
  The investigators plan to prospectively collect data and monitor the outcome of each hip patient. Subjects will complete a number of assessments utilizing iPads with an electronic data collection system. The data will be collected during each visit or done remotely via the internet, at which time the adjusted means from this longitudinal model will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: James Genuario, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided